CLINICAL TRIAL: NCT00330551
Title: Effects of Risperdal Consta Versus Oral Antipsychotic Medication on Clinical and Functional Outcome and Neurocognition in First-episode Schizophrenia
Brief Title: Oral Versus Injectable Risperidone for Treating First-Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Keith Nuechterlein, Ph.D., Professor, University of California, Los Angeles, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P50MH066286 (NIH); P50MH066286 (NIH); DATR A2-AISZ (Registry Identifier: World Health Organization ICTRP); Janssen RIS-NAP-4009 (Other Grant/Funding Number: Janssen Scientific Affairs)
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2020-03-23 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Schizophrenia
Keywords: Schizoaffective Disorder, Depressed Type; Schizophreniform Disorder; First-episode Schizophrenia; Injectable Risperidone
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Long-acting injectible risperidone (Experimental): Participants who are randomly assigned to this arm will be administered the long-acting injectible form of risperidone (Risperdal Consta) every two weeks, plus group skills training and case management, for 12 months.
  Interventions: Drug: Risperidone in Long-Acting Injectable Form (Consta)
- Oral risperidone (Active Comparator): Participants who are randomly assigned to this arm will be treated with the oral version of risperidone (Risperdal) daily, plus group skills training and case management, for 12 months.
  Interventions: Drug: Oral Risperidone

INTERVENTIONS:
Drug: Oral Risperidone — Patients will be treated with oral risperidone daily, with the dosage determined by treating psychiatrist.
  Other Names: Risperdal
  Arms: Oral risperidone
Drug: Risperidone in Long-Acting Injectable Form (Consta) — Participants will take a 25 mg dosage of injectable risperidone (Risperidone in Long-Acting Injectable Form (Consta)) once every 2 weeks. Dosage will be adjusted if needed.
  Other Names: Risperdal Consta
  Arms: Long-acting injectible risperidone

SUMMARY:
This study will determine the effectiveness of oral risperidone versus long-acting injectable risperidone in treating people with first-episode schizophrenia.

DETAILED DESCRIPTION:
Schizophrenia is a severely disabling brain disorder. People with schizophrenia often experience hallucinations, delusions, thought disorders, and movement disorders. Proper treatment of first-episode schizophrenia may increase the chances of controlling disease progression on a long-term basis. People experiencing their first episode of schizophrenia are more responsive to treatment than those with chronic schizophrenia, but are also more susceptible to adverse treatment side effects. Atypical antipsychotic medications have been shown to produce fewer adverse side effects than older "typical" antipsychotics. Risperidone is a type of atypical antipsychotic medication that is used to control the symptoms of schizophrenia. This study will determine the effectiveness of oral risperidone versus long-acting injectable risperidone in treating people with first-episode schizophrenia.

Participants in this open label study will be randomly assigned to receive either orally administered risperidone or long-acting risperidone administered via injection. Participants assigned to oral risperidone will receive medication in doses that are determined to be optimal by the study psychiatrist. Participants assigned to long-acting risperidone will receive an injection of risperidone once every 2 weeks. Dosages will begin at 25 mg and will be adjusted as necessary to achieve the optimal dosage. Following 2 to 3 months to achieve outpatient risperidone dosage stabilization, the randomized medication conditions will begin and participants will be monitored for 1 year. Study visits will occur once weekly throughout the study. They will include group therapy meetings focused on everyday living skills; family education about schizophrenia; assessments of medication response; and individual meetings with a case manager for counseling and evaluations of schizophrenia symptoms.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia, schizoaffective disorder (depressed type), or schizophreniform disorder
* First major episode of psychotic symptoms occurred within 2 years prior to study entry
* Participant in the UCLA Center for Neurocognition and Emotion in Schizophrenia

Exclusion Criteria:

* Neurological disorder or injury (e.g., encephalitis, epilepsy, traumatic brain injury)
* Mental retardation (e.g., premorbid IQ less than 70)
* Significant alcohol or substance abuse within 6 months prior to study entry
* Inability to complete research measures in English
* Any condition that may make risperidone use medically inadvisable

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 126 (Actual)
Dates: Start 2006-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith H. Nuechterlein, PhD, Principal Investigator — University of California, Los Angeles, Department of Psychiatry and Biobehavioral Sciences
Locations (1):
- Semel Institute for Neuroscience and Human Behavior at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Subotnik KL, Casaus LR, Ventura J, Luo JS, Hellemann GS, Gretchen-Doorly D, Marder S, Nuechterlein KH. Long-Acting Injectable Risperidone for Relapse Prevention and Control of Breakthrough Symptoms After a Recent First Episode of Schizophrenia. A Randomized Clinical Trial. JAMA Psychiatry. 2015 Aug;72(8):822-9. doi: 10.1001/jamapsychiatry.2015.0270. PMID 26107752
- [Derived] Bartzokis G, Lu PH, Amar CP, Raven EP, Detore NR, Altshuler LL, Mintz J, Ventura J, Casaus LR, Luo JS, Subotnik KL, Nuechterlein KH. Long acting injection versus oral risperidone in first-episode schizophrenia: differential impact on white matter myelination trajectory. Schizophr Res. 2011 Oct;132(1):35-41. doi: 10.1016/j.schres.2011.06.029. Epub 2011 Jul 20. PMID 21767934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 126 eligible and enrolled participants, 43 dropped out prior to the start of randomized treatment, resulting in 83 randomized.
Groups:
- Long-acting Injectable Risperidone: Participants taking risperidone, administered in injectable long-acting form (Risperdal Consta), plus group skills training and case management
  Group Skills Training and Psychoeducation: Group skills training sessions will be weekly throughout the study. The sessions will include group therapy meetings focused on everyday living skills, family education about schizophrenia, assessments of medication response, and individual meetings with a case manager for counseling and evaluations of schizophrenia symptoms.
  Individual Case Management: An individual therapist will provide therapy focused on everyday life skills and aid in interfacing with community agencies, work, and/or school settings.
  Risperidone in Long-Acting Injectable Form (Consta): Participants will take a 25 mg dosage of injectable risperidone once every 2 weeks. Dosage will be adjusted if needed.
- Oral Risperidone: Participants taking daily oral risperidone, plus group skills training and case management
  Group Skills Training and Psychoeducation: Group skills training sessions will be weekly throughout the study. The sessions will include group therapy meetings focused on everyday living skills, family education about schizophrenia, assessments of medication response, and individual meetings with a case manager for counseling and evaluations of schizophrenia symptoms.
  Individual Case Management: An individual therapist will provide therapy focused on everyday life skills and aid in interfacing with community agencies, work, and/or school settings.
  Oral Risperidone: Daily oral risperidone dosage will determined by treating psychiatrist.
Period: Overall Study
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Started | 40 | 43
Completed | 30 | 27
Not Completed | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone | Total
Number analyzed (Participants) | 40 | 43 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 9 | 12
  Between 18 and 65 years | 37 | 34 | 71
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.9 (3.8) | 21.1 (3.2) | 21.5 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 31 | 34 | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 20 | 35
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 14 | 9 | 23
  White | 18 | 23 | 41
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 43 | 83

OUTCOME MEASURES:

1. Primary Outcome: Medication Adherence
Description: 5-point scale (1 = best adherence, 5= nonadherent) based on pill counts, MEMS cap readings, plasma assays, and psychiatrist judgments for oral risperidone and timing of injections for long-acting injectable risperidone averaged over study participation
Time Frame: Measured weekly throughout study participation, averaged over study participation
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Long-acting Injectable Risperidone: Participants who are randomly assigned to this arm will be administered the long-acting injectable form of risperidone (Risperdal Consta) every two weeks, plus group skills training and case management, for 12 months.
  Risperidone in Long-Acting Injectable Form (Consta): Participants will take a 25 mg dosage of injectable risperidone (Risperidone in Long-Acting Injectable Form (Consta)) once every 2 weeks. Dosage will be adjusted if needed.
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 40 | 43
units on a scale | 1.1 (0.5) | 1.9 (0.8)
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p = .05, t-test, 2 sided; t-test = .77, 95% CI 2-sided [0.483 to 1.058]; t(80)=5.3, p<.001

2. Primary Outcome: Number of Participants Who Had an Exacerbation or Relapse of Psychotic Symptoms
Description: Dichotomous measure: Presence of any of three psychotic relapse or exacerbation categories scored from the Brief Psychiatric Rating Scale (BPRS) occurring any time after randomization and until end of study participation (up to 12 mos.).
Time Frame: Occurrence after randomization and until end of study participation (up to 12 mos.)
Population: All participants randomized to long-acting injectable or oral risperidone
Measure: Count of Participants; unit: Participants
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 40 | 43
Participants | 2 | 14
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p = .001, Chi-squared; Risk Difference (RD) = 11.1

3. Primary Outcome: Number of Participants Who Returned to Work or School (SAS Work Section)
Description: The Social Adjustment Scale records the return to work or school and the number of weeks in work or school during each 3-month period. For this outcome, outcome as dichotomized as 0 if an individual did not return to work or school and 1 if they did return to competitive work or regular school enrollment.
Time Frame: Measured from Baseline to Month 12
Population: All participants with data regarding return to work or school
Measure: Count of Participants; unit: Participants
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 37 | 38
Participants | 29 | 29
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p = .83, Chi-squared

4. Primary Outcome: Number of Weeks Maintaining Work or School (SAS)
Description: Measured as the number of weeks in which a participant has competitive employment or attends regular school courses. Possible range is 0 to 52 weeks.
Time Frame: Cumulative total measured from Baseline to Month 12
Population: All participants with data on duration of work or school
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 37 | 41
weeks | 26.7 (20.4) | 21.1 (18.0)
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; A priori hypothesis was that long-acting injectible risperidone would lead to greater duration of work/school attendance than oral risperidone; Test type: Superiority; p = .20, ANOVA

5. Primary Outcome: Change in Global Functioning Scale: Role
Description: 10-point scale of work/school functioning. Scale range is from 1 (extreme role dysfunction) to 10 (superior role functioning). Measured by subtracting the baseline rating from the rating at 12 months.
Time Frame: Measured at Baseline and Month 12
Population: All participants with Global Functioning Scale: Role ratings at baseline and 12 months
Measure: Mean (Standard Deviation); unit: Changes on a 10-point scale
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 29 | 30
Changes on a 10-point scale | 1.5 (2.7) | 1.2 (3.0)
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p = .71, ANOVA

6. Secondary Outcome: MATRICS Consensus Cognitive Battery (MCCB) Overall Composite T Score
Description: The MCCB Overall Composite T score is computed by the MCCB Computer Scoring Program from the raw scores for 10 individual cognitive tests. The mean for the general population of comparable age and sex is 50 with a standard deviation of 10. Higher scores indicate better cognitive functioning. The outcome measure was the change from baseline to 12 months, calculated as 12-month T score minus baseline T score. Higher values indicate better outcome.
Time Frame: Measured at baseline and 12 months
Population: All participants with MCCB Overall Composite scores at baseline and 12 months
Measure: Mean (Standard Deviation); unit: Change score: change in T scores
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 29 | 32
Change score: change in T scores | 3.5 (7.5) | 4.4 (5.0)
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p = .57, ANOVA

7. Secondary Outcome: Emotional Reactivity on Psychophysiological Measures
Description: Electrodermal reactivity to pictures of negative versus neutral stimuli was the initially proposed measure. Larger skin conductance increases in response to negative pictures compared to neutral pictures would indicate stronger emotional reactivity.
Time Frame: Measured from Baseline to Month 12
Population: No data were available because this part of the initial proposal was not funded.
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Retention in Treatment
Description: Number of days on the randomized medication before being switched to a different antipsychotic medication or dropping out of the medication trial. Possible range is 0 to 365, with higher numbers indicating better retention in treatment.
Time Frame: From baseline to 12 months
Population: All participants randomized to oral vs. long-acting injectable risperidone
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 40 | 43
days | 307.6 (108.3) | 270.7 (126.4)
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p < .16, ANOVA

9. Secondary Outcome: Awareness of Illness, as Assessed by the Scale to Assess Unawareness of Mental Disorder-Revised (SUMD-R)
Description: Rating scale based on clinician's interview of patient to determine level of lack of awareness of having a mental disorder. Range is from 1 (Aware) to 5 (Unaware), so lower scores indicate better outcome.
Time Frame: Baseline to 12 months
Population: All participants with ratings at baseline and 12 months, with 6-month rating carried forward if no 12-month rating was completed.
Measure: Mean (Standard Deviation); unit: Change scores on 5-point rating scale
Arm/Group | Long-acting Injectable Risperidone | Oral Risperidone
Number analyzed (Participants) | 30 | 34
Change scores on 5-point rating scale | .07 (1.34) | -.24 (1.56)
Statistical Analysis 1: Comparison: Long-acting Injectable Risperidone vs Oral Risperidone; Test type: Superiority; p = .41, ANOVA

ADVERSE EVENTS:
Groups:
- Long-acting Injectible Risperidone: Participants taking risperidone, administered in injectible long-acting form (Risperdal Consta), plus group skills training and case management
  Group Skills Training and Psychoeducation: Group skills training sessions will be weekly throughout the study. The sessions will include group therapy meetings focused on everyday living skills, family education about schizophrenia, assessments of medication response, and individual meetings with a case manager for counseling and evaluations of schizophrenia symptoms.
  Individual Case Management: An individual therapist will provide therapy focused on everyday life skills and aid in interfacing with community agencies, work, and/or school settings.
  Risperidone in Long-Acting Injectable Form (Consta): Participants will take a 25 mg dosage of injectable risperidone once every 2 weeks. Dosage will be adjusted if needed.
Arm/Group | Long-acting Injectible Risperidone | Oral Risperidone
Serious Adverse Events (participants affected / at risk) | 2/40 | 8/43
Other Adverse Events (participants affected / at risk) | 11/40 | 19/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long-acting Injectible Risperidone (N=40) | Oral Risperidone (N=43)
psychiatric hospitalization (Psychiatric disorders) | 2 (2) | 8 (8) — psychiatric hospitalization
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Long-acting Injectible Risperidone (N=40) | Oral Risperidone (N=43)
BMI increase from normal or overweight to Obese (Metabolism and nutrition disorders) | 7 (7) | 5 (5) — increase in BMI from normal or overweight to any Obese category
Lipid Increase (Vascular disorders) | 2 (2) | 9 (9) — Increase in LDL or Triglycerides from normal to high
Tardive Dyskinesia (Nervous system disorders) | 2 (2) | 3 (3) — New onset of mild symptoms of Tardive Dyskinesia
Prolactin related (Endocrine disorders) | 3 (3) | 4 (4) — Symptoms related to prolactin levels

LIMITATIONS AND CAVEATS:
This trial used oral risperidone as the comparator to allow a strong comparison between oral and long-acting injectable forms of the same drug. Generalization of results to other oral antipsychotic medications was not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No